CLINICAL TRIAL: NCT06042582
Title: From Nature to Bedside- Algae Based Bio Compound for Prevention and Treatment of Inflammation, Pain and IBD
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Silvio Danese, Director of Gastroenterology and Endoscopy Unit, IRCCS San Raffaele
Other Study IDs: Algae4IBD
Record Dates: First submitted 2023-08-29; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: IBD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ulcerative Colitis (UC): * subjects undergoing endoscopy and biopsies collection per standard of care
  * adult patients ≥18 and <60 years
  * clinical and endoscopic evaluation (Mayo score≥2)
  Interventions: Procedure: Additional biopsies collection
- Crohn's Disease (CD): * subjects undergoing endoscopy and biopsies collection per standard of care
  * adult patients ≥18 and <60 years
  * clinical and endoscopic evaluation (Harvey-Bradshaw score ≥5 and overall simplified endoscopic score (SES-CD) >2)
  Interventions: Procedure: Additional biopsies collection
- NO UC/CD: * subjects undergoing endoscopy and biopsies collection (≥18 and <60 years) according to the normal clinical practice (as patients undergoing cancer surveillance, irritable bowel syndrome (IBS), diarrhea)
  * subjects not affected by UC or CD according to the previously reported clinical and endoscopic evaluation criteria
  Interventions: Procedure: Additional biopsies collection

INTERVENTIONS:
Procedure: Additional biopsies collection — We will recruit only subjects (UC, CD and NO-UC/CD) scheduled for the endoscopy and biopsies-collection according to the usual clinical practice. During the endoscopy we will collect 6 additional biopsies.

SUMMARY:
This study is part of the project funded by the Horizon2020 program for establishing the consortium Algae4IBD (https://algae4ibd.eu/), where OSR participates as a partner. It aims to promote the implementation of the European Crohn's and Colitis Organization (ECCO/FECCO) Directive and the benefit of the Inflammatory Bowel Disease (IBD) patient's wellness by finding innovative algae based novel small molecule therapeutics. A systemic approach to eco-innovation is adopted to create interconnections between sectors, value chains, natural resources, and relevant societal stewards. To this end, the consortium has set specific objectives to achieve holistic innovations, including technical, economic, health, and social factors that all work in concert.

IBD included Crohn's disease and ulcerative colitis. It is a class of chronic inflammatory disorders with complex pathogenesis. Despite the lack of a full understanding of its etiogenesis, many anti-inflammatory treatments have been developed over the last decades. However, not all patients may benefit from these treatments and some of them are refractory to the current therapies or experience relapse of the disease. Therefore, there is still an urgent need to find an innovative line of interventions for ameliorating these patients' overall quality of life.

Algae4IBD consortium will form a bridge between innovation and market demands to prevent and treat inflammation, pain, and IBD. Bioactive molecule/compounds extracts from microalgae, cyanobacteria, and macro-algae (MiaCyMa) are an inexhaustible untapped natural source for products destined for IBD prevention and treatment (inflammation, pain, and the disease process associated with the gut's microbiome). The natural source potential is still more promising when considering extremophile strains for excellent metabolism systems. Moreover, the production of the natural source of biological materials should be sustainable. Indeed, the non-genetically modified organisms (GMO cultures offer numerous advantages such as reduced requirements of fresh water and land (no arable land is required), drastic reduction of nitrogen sources, and potential environmental threats. Algae4IBD concept will include a multi-step screening approach and feedback loops across the project steps to achieve its goals. Specifically, OSR is in charge with work package (WP) 4, task 4.4, which aims to characterize the activity of plant cell (algae) extracts named in this proposal as "natural compounds" of algae provided by the consortium in ex-vivo models, using bioptic samples derived from patients with IBD (patients with ulcerative colitis (UC) and Crohn's disease (CD)), comparing them to samples derived from patients without UC and CD.

ELIGIBILITY:
INCLUSION CRITERIA

SUBJECTS WITH THE DIAGNOSIS OF UC OR CD:

* subjects undergoing endoscopy and biopsies collection per standard of care
* adult patients ≥18 and <60 years

Additionally, for people with UC:

- clinical and endoscopic evaluation (Mayo score≥2)

Additionally, for individuals with CD:

- clinical and endoscopic evaluation (Harvey-Bradshaw score ≥5 and overall simplified endoscopic score (SES-CD) >2)

SUBJECTS NOT AFFECTED BY UC OR CD:

* subjects undergoing endoscopy and biopsies collection (≥18 and <60 years) according to the normal clinical practice (as patients undergoing cancer surveillance, irritable bowel syndrome (IBS), diarrhea)
* subjects not affected by UC or CD according to the previously reported clinical and endoscopic evaluation criteria All patients will sign the informed consent.

EXCLUSION CRITERIA

SUBJECTS WITH THE DIAGNOSIS OF UC OR CD:

- subjects with UC or CD who do not have the previously described clinical and endoscopic evaluation criteria

SUBJECTS NOT AFFECTED BY UC OR CD (CONTROL GROUP):

-subjects undergoing anti-inflammatory and/or immunosuppressive treatments for other diseases not related to UC or CD

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will recruit adult patients with CD or UC and without CD and UC, ≥18 and <60 years and without any previously documented gastrointestinal infections in collaboration with the Gastroenterology and Digestive Endoscopy unit (IRCSS Ospedale San Raffaele). CD and UC diagnosis will be determined by clinical and endoscopic scores (described below in inclusion criteria). Control data will come from the same intestinal areas of age-matched no-UC/CD subjects undergoing endoscopic surveillance for not IBD-related conditions (described into the inclusion criteria) according to the standard of care.
  The participation is voluntary and the patient is allowed to refuse further participation in the protocol whenever he/she wants.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the response of intestinal mucosa samples to treatments with natural compounds derived from algae in terms of release of pro-inflammatory factors (1), transcriptomics, metatranscriptomics (2) and lipidomics analysis (3) | 30 months
  1. Release of pro-inflammatory cytokines using ELISA
  2. RNA-Seq-generated FASTQ reads from human colons will be quality filtered and adaptor trimmed with NCBI fastq-dump.
  3. Lipids detected by LC-MS/MS will be classified based on their precursors, and, in parallel, based on their metabolic pathways.
  By multi-omic factor analysis we will integrate these data with the patients' clinical parameters, correlating among each other in parallel and giving one single output (outcome measure, in our case, multiomic factor) explaining how the different omic layers are assigned simultaneously to specific clinical characteristics, thus resulting as associated with, or predictive of, the clinical progression of IBD.

IPD SHARING:
Plan to Share IPD: Undecided